CLINICAL TRIAL: NCT04089046
Title: Telemedicine Enhanced Asthma Management - Uniting Providers for Teens
Brief Title: Telemedicine Enhanced Asthma Management - Uniting Providers for Teens (TEAM-UP for Teens)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Johns Hopkins University (Other); University of Arkansas (Other)
Responsible Party: Principal Investigator, Jill Halterman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00004160
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAM-UP for Teens Intervention (Experimental): TEAM-UP for Teens pairs school-based and video-supported directly observed therapy (DOT) of daily preventive asthma medications with specialist care and ongoing self-management support using live, real-time telemedicine through school.
  Interventions: Behavioral: TEAM-UP for Teens
- Enhanced Care Comparison (Active Comparator): Teens in the EC group will receive a symptom assessment and asthma education materials at baseline, and their PCPs will be contacted by facsimile or email to recommend DOT of preventive asthma medication through school as well as referral to an asthma specialist. Systematic reminders will be sent to the family and PCPs to schedule recommended healthcare visits and consider specialist referral at the same intervals as the TEAM-UP group's virtual visits.
  Interventions: Behavioral: Enhanced Care (EC)

INTERVENTIONS:
Behavioral: TEAM-UP for Teens — TEAM-UP for Teens pairs school-based directly observed therapy (DOT) of daily preventive asthma medications with specialist care and ongoing self-management support using live, real-time telemedicine through school.
  Arms: TEAM-UP for Teens Intervention
Behavioral: Enhanced Care (EC) — Teens in the EC group will receive a symptom assessment and asthma education materials at baseline, and their PCPs will be contacted by facsimile or email to recommend DOT of preventive asthma medication through school as well as referral to an asthma specialist. Systematic reminders will be sent to the family and PCPs to schedule recommended healthcare visits and consider specialist referral at the same intervals as the TEAM-UP group's virtual visits.
  Arms: Enhanced Care Comparison

SUMMARY:
Low-income, minority teenagers have disproportionately high rates of asthma morbidity, including excess risk of emergency department visits, hospitalizations, and death from asthma. Despite well established guidelines, under-treatment for asthma is common, particularly for poor urban teens. This study aims to test a novel, developmentally appropriate and scalable model of care to ensure optimal guideline-based treatment for urban teens with difficult to control asthma. The Telemedicine Enhanced Asthma Management-Uniting Providers for Teens (TEAM-UP for Teens) program includes 3 core components: 1- An individualized asthma management plan developed at the start of the school year via a real-time, synchronous school-based telemedicine visit that directly connects the teen to an asthma specialist, 2- School-based or video supported directly observed therapy (DOT) to implement the medication plan and allow for teens to experience the benefits of consistent therapy, 3- Follow-up telehealth visits with a nurse asthma educator to facilitate ongoing care and provide developmentally appropriate self-management support. This study is a randomized trial of TEAM-UP for Teens vs an enhanced care (EC) control group (n=360, 12-16 years). We will assess the effectiveness of the program in reducing morbidity and improving guideline-based asthma care. Our main hypothesis is that Teens receiving the TEAM-UP for Teens intervention will have more symptom-free days at 3, 5, 7, and 12-months compared to EC. We will assess a number of secondary outcomes, including additional clinical outcomes, functional outcomes, airway inflammation, and receipt of specific care measures including medication adjustments and treatment of and other comorbidities. We will also identify potential mediators and moderators of the intervention effect, and will evaluate the process of intervention implementation. At the completion of the study, the program will be better defined as a sustainable means to improve care and reduce morbidity for high risk teens with difficult to control asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-diagnosed asthma (based on caregiver report with validation from teen's physician).
2. Moderate-severe persistent severity (requiring Step 3 or higher care) or asthma that is uncontrolled despite therapy
3. Age >=12 and =<17 years
4. Residence in the City of Rochester and surrounding metro area.

Exclusion Criteria:

1. Inability to speak and understand either English or Spanish. (*Participants unable to read will be eligible, and all instruments will be given verbally.)
2. Current participation in an asthma study
3. Planning to move outside of Rochester in less than 6 months
4. If they have received asthma specialist care in the prior 3 months, they will be asked if they would be comfortable seeing an additional asthma specialist for our study if their current specialist is unable to participate in the study. If the family is not comfortable with seeing an additional asthma specialist for the study, they will be excluded.
5. Having other significant medical conditions (congenital heart disease, cystic fibrosis, other chronic lung disease) that could interfere with the assessment of asthma-related measures
6. In foster care or other situations in which consent cannot be obtained from a guardian

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Symptom Free Days in prior 14 days | 12-month
  Mean Symptom Free Days will be calculated as a mean using data collected at 3-, 5-, 7- and 12-months post baseline. Caregivers and teens will report the number of days the teen experienced no symptoms of asthma (defined as 24 hrs with no coughing, wheezing, shortness of breath, and no need for rescue medicine) in the past 2 weeks (range 0-14).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sets to be submitted to the NHLBI Data Repository will include baseline, follow up visit, procedural based data, and outcome data. Prior to providing data, patient identifiers will be deleted, original identification numbers will be replaced with new, randomized identification numbers, dates will be coded relative to date of enrollment, and identifiers will be removed. Variables such as socioeconomic and demographic data, household and family composition, anthropometric measures, prior medical conditions, and parent and teen medical history will be grouped or recoded.